CLINICAL TRIAL: NCT06354569
Title: Risk Factors and Risk Grading Prediction of Perioperative Respiratory Adverse Events in Children
Status: Recruiting | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yanyu Liu, Principal Investigator, Sichuan Provincial People's Hospital
Other Study IDs: 2022.232
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Perioperative Respiratory Adverse Events
Keywords: respiratory adverse events, risk prediction, children

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
to explore the risk factors of perioperative respiratory adverse events in children, and to establish a risk prediction model of perioperative respiratory adverse events in children

DETAILED DESCRIPTION:
600 children undergoing elective surgery under general anesthesia were selected. Age, sex, weight, height, allergy history, past history, snoring, passive smoking, abnormal laboratory examination and chest X-ray before operation, upper respiratory tract infection 14 days before operation, Operation Site, working years of anesthesiologist, anesthesia method, Operation Duration, anesthesia duration, perioperative vital signs and respiratory adverse events were collected. The risk prediction model of perioperative respiratory adverse events in children was established by using LASSO (least absolute shrinkage and selection operator) algorithm and gradient boosting machine (GBM) algorithm to screen the relevant data collected during routine diagnosis and treatment, such as demographic characteristics, physical conditions, airway sensitivity, environmental sensitivity and anesthesia management

ELIGIBILITY:
Inclusion Criteria:

* （1）Children aged 1 month to 12 years, （2） ASA Class I or II, （3）scheduled for surgery under general anesthesia

Exclusion Criteria:

-（1）Children and guardians declined to participate in the study (2) children with severe chronic respiratory, cardiovascular, central nervous system, liver and kidney diseases; (3) on the day of operation, the patients had active URTI and pulmonary infection, such as severe nasal obstruction, large amount of airway secretion, severe cough, fever (body temperature > 37.5 ° C) , in addition to the above symptoms, signs of pulmonary consolidation and/or wet Rales, or peripheral white blood cells > 10 × 109/L or < 4 × 109/L with or without left shift of the nucleus, and chest X-ray showed new patchy, patchy infiltrative shadows or interstitial changes.

(4) the child had severe anaphylaxis to narcotic drugs

Ages: 1 Month to 12 Years | Sex: All
Age Groups: Child
Study Population: Children aged 1 month to 12 years, Asa Class I or II, scheduled for surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of perioperative respiratory adverse events | perioperative
  Collection of respiratory adverse events including laryngeal spasm, Bronchospasm, decreased oxygen saturation, and increased secretions

CONTACTS AND LOCATIONS:
Overall Officials: Ting Xu, Study Director — Sichuan provincial Peopel'Hospital
Locations (1):
- Sichuan provincial Peopel'Hospital, Chengdu, Sichuan, China